CLINICAL TRIAL: NCT05253560
Title: Prodromal Parkinsonian Features in GBA1 Mutation Carriers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Ari Zimran, Prof., Shaare Zedek Medical Center
Other Study IDs: SZMC-0168-17
Record Dates: First submitted 2021-11-11; First posted 2022-02-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Gaucher Disease, Type 1; Healthy
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample for DNA sequencing and biomarker analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Carriers of Gaucher disease: Family of patients with Gaucher disease, sequenced for the GBA1 gene.
  Interventions: Diagnostic Test: The investigators aim to identify prodromal PD in a cohort of carriers of Gaucher disease.
- Gaucher patients: Patients from the Gaucher clinic in Shaare Zedek Medical Center, Jerusalem, Israel
  Interventions: Diagnostic Test: The investigators aim to identify prodromal PD in a cohort of carriers of Gaucher disease.
- Healthy controls: Family members of Gaucher patients who are not carriers of Gaucher disease
  Interventions: Diagnostic Test: The investigators aim to identify prodromal PD in a cohort of carriers of Gaucher disease.

INTERVENTIONS:
Diagnostic Test: The investigators aim to identify prodromal PD in a cohort of carriers of Gaucher disease. — Tests to help identify prodromal PD in a cohort of carriers of Gaucher disease

SUMMARY:
Objective of the trial. To define a sub-population which is at increased risk of developing Parkinson, beyond the fact of carrying Gaucher; in this sub-population the investigators shall conduct a comprehensive evaluation that includes a variety of non-invasive tests, whose purpose is to evaluate the state of the pre- Parkinson's disease signs, signs which can appear, even twenty years before the appearance of the disease, and also to compare them to a group of diagnosed Gaucher patients and a group of healthy people who are not carriers of Gaucher disease.

A group of those carriers will be available for trial or for treatment, if there will be a medicine for the prevention of the development of Parkinson, obtainable.

DETAILED DESCRIPTION:
The carriers, the healthy people and the Gaucher patients will undergo a number of non-invasive tests, which test the pre-Parkinson signs.

The tests are based on various sense tests, blood tests, measuring of blood pressure, lying and standing, ultra-sound of the brain and a neurological test (test of the nervous system and various questionnaires).

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate

Exclusion Criteria:

* PD patients
* Dementia

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Carriers of Gaucher disease mutation Gaucher patients Healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-05-16 (Actual); Primary Completion 2024-01-16 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Building a model to identify carriers of Gaucher disease prone to Parkinson's disease, using tests to assess different domains of PD, including anatomy, cognitive and mental, sleep disorder, and motor. | 8 Years
  Carriers of a variant in the GBA1 gene (GBA carriers) are at the highest risk of developing Parkinson disease (PD). A screening study for prodromal PD features in a cohort of obligatory GBA carriers between 40-75 years was initiated to identify candidates for a PD prevention trial. We added healthy controls and GD patients in order to determine the incidence of prodromal PD and for analyzing the differences between the two groups helping to build a model for identifying at risk PD at the prodromal stage.
  Participants preform 15 pre-defined non-invasive tests for prodromal PD and assessment of risk factors. Risk factors for PD included age, sex, type of GBA1 variant, coffee and tea caffeine consumption, smoking habits, exposure to solvents and pesticides, and family history of PD (1st and/or 2nd degree relatives with PD).

OTHER OUTCOMES:
Transcranial sonography (TCS) | 8 years
  Transcranial sonography (TCS) is a useful noninvasive diagnostic tool to detect hyperechogenicity (SN+) of the substantia nigra area in the brain. The hyperechogenicity happens due to increased amounts of iron, reflecting a functional impairment.
Color discrimination test | 8 years
  Color discrimination was analyzed using The Farnsworth-Munsell 100 hue test. The test includes four boxes with a fixed number of color shade caps with slight shade differences needed to be ordered correctly. The result of each box was entered into a computerized system and automated the total error score (TES)
Hyposmia by the Bit-A UPSIT smell test | 8 years
  The shorter version of the UPSIT smell test (The University of Pennsylvania Smell Identification Test) was used to evaluate hyposmia using twelve cards, each with a different smell.
Orthostatic hypotension (OH) | 8 years
  defined as a fall of at least 20 mmHg systolic or at least ten mmHg diastolic blood pressure by 3 min of active standing or head-up tilt
Montreal Cognitive Assessment (MoCA) | 8 years
  evaluate the cognitive and mental aspects associated with PD. A Montreal Cognitive Assessment (MoCA) score of 26 and above was considered normal
NeuroTrax computerized battery. | 8 years
  The NeuroTrax computerized battery (www.neurotrax.com) includes seven sections: memory, executive function, attention, information processing speed, visual-spatial, verbal function, and motor skills
Beck Depression Inventory | 8 years
  self-administered questioner including 21 questions used to screen, diagnose, and measure the severity of depression.
Frontal lobe assessment battery (FAB). | 8 years
  evaluates executive dysfunction
rapid eye movement (REM) | 8 years
  Idiopathic rapid eye movement sleep behavior disorder is an important risk factor in the diagnosis of PD. The REM questionnaire was completed by the participant.
Epworth sleepiness scale (ESS) | 8 years
  assessing daytime sleepiness includes an eight-question questionnaire scoring between 0 and 24; the higher the score, the higher the chances of dosing off
Perdue pegboard. | 8 years
  Perdue pegboard measures the movement of fingers, hands, and arms in 4 different tasks, testing motor abilities and coordination by placing as many pegs and discs on a board in three 30 seconds trials for each subset and three 60 second trials for the assembly subset
UPDRS part III. | 8 years
  measures gross motor function. A score above 6, not including postural and action tremor, was considered abnormal
The Timed Up and Go (iTUG). | 8 years
  The Timed Up and Go (iTUG) (EncephaLogTM) is a platform that utilizes smartphones' internal motion sensors for conducting motor evaluation including general walking score, step to step persistency, hand sway and rotation time.
Questionnaire regarding risk factors | 8 years
  Spontaneous bowel movement frequency was used to define constipation. Urinary and erectile dysfunction were assessed according to the MDS criteria

CONTACTS AND LOCATIONS:
Overall Officials: Ari Zimran, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Michal Becker- Cohen, Jerusalem, Please Select..., Israel

IPD SHARING:
Plan to Share IPD: Undecided